CLINICAL TRIAL: NCT05149092
Title: Randomized, Double Blind, Placebo Controlled Study to Investigate the Effect of Chicken Protein Hydrolysates (CPH) in Persons With High Waist Circumference
Brief Title: Effects of Chicken Protein Hydrolysate (CPH) Supplementation in People With High Waist Circumference
Acronym: CHICKPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Norilia AS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPH-Study
Record Dates: First submitted 2021-03-09; First posted 2021-12-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Abdominal Obesity
Keywords: Cardiovascular disease risk; Protein supplementation; Metabolic health
MeSH Terms: conditions — Obesity, Abdominal | interventions — Caseins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (casein protein supplement) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Chicken protein hydrolysate supplement (Active Comparator)
  Interventions: Dietary Supplement: Chicken protein hydrolysate supplement

INTERVENTIONS:
Dietary Supplement: Chicken protein hydrolysate supplement — Daily oral self-administration of 18 g of supplement dissolved in water/mineral water, spread over 2-3 occasions
  Other Names: CPH
  Arms: Chicken protein hydrolysate supplement
Dietary Supplement: Placebo — Daily oral self-administration of 18 g of supplement dissolved in water/mineral water, spread over 2-3 occasions
  Other Names: Casein
  Arms: Placebo (casein protein supplement)

SUMMARY:
In this randomized, placebo controlled, double blind trial, effects of relatively high doses of chicken protein hydrolysate (CPH) or casein hydrolysate (placebo) supplementation will be investigate in healthy persons with abdominal obesity. The 12-week study examines potential effects on body weight, abdominal obesity, body composition, plasma parameters of metabolic health including lipids, inflammatory parameters, redox state and microbiota biomarkers.

DETAILED DESCRIPTION:
Small peptides in the range of 2 - 12 amino acids are believed to cross the intestinal wall undigested and enter the circulation where they can have a range of activities based on their amino acid composition and structure. Natural peptides isolated from a number of food proteins, including plants and marine organisms, are shown to have antioxidant effects in in vitro tests, and anti-hypertensive effects in mice through inhibition of the angiotensin-converting-enzyme (ACE). Protein hydrolysates from both animal- and plant-based sources will consist of a mixture of potentially bioactive peptides that can have specific effects based on their composition. Studies have shown that egg- and soy-derived hydrolysates have anti-diabetic and anti-obesity properties in rodents. Pre-clinical studies in mice have demonstrated potent plasma cytokine lowering abilities and atherosclerosis-prevention by chicken protein hydrolysate (CPH) diets, as well as effects on plasma cholesterol level, cytokines and lipid metabolism, including mitochondrial function. In addition, an isolated peptide fraction from chicken inhibits the dipeptyl peptidase IV, and thus has the potential to restore glucose homeostasis in type 2 diabetics.

The hydrolysate supplements used in this study are obtained from rest raw materials (RRM) from mechanical deboning of chicken meat (Food Grade, Nortura AS Hærland, Norway). Freshly minced chicken RRM has been treated with enzymes optimized to generate bioactive hydrolysates. The supplement is given in a dose of 18 g protein per day, corresponding to the protein content of a standard meal, and similar to doses recommended in protein shake supplements.

Around 60 males and females age >20 years with abdominal obesity participate, recruited primarily through social media advertisements (Facebook) limited to a 12 km radius around the city center of Bergen. Participants provided written informed consent, and were screened via self-reporting in an online form in EasyTrial hosted by the Research Unit for Clinical Trials at the University of Bergen. Data collection by the study staff at baseline verifies inclusion and exclusion criteria and participant eligibility prior to randomization. The potential participants are informed about practical details at a digital or physical meeting 1-2 weeks prior to baseline.

Groups of participants (40-60% males/females) are block randomized to the two treatments (CPH or placebo casein supplementation) using randomly selected block sizes, and stratified according to sex.

The participants are given a container with the powder sufficient for the entire 12-week study period, and a spoon to measure the intake at breakfast (6 g), lunch (6 g) and supper (6 g), or morning (9 g) and evening (9 g) according to individual preference. The patients will mix the powder products in water or mineral water.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects at least 20 years old understanding Norwegian oral and written information
* Waist circumference of:

  * Men > 95 cm
  * Women > 81 cm

Exclusion Criteria:

* Pregnancy
* Having used high-dose omega-3 PUFA supplements (>2 g/day) 28 days' prior to randomization
* Alcohol or drug abuse or any conditions associated with poor compliance
* Scheduled hospitalization during the course of the study that could compromise the study
* Major diseases or infections including chronic diseases
* Known or suspected sensitivity or allergic reactions to the IMP or excipients
* Presence of other major medical or psychiatric illness that would affect the ability to participate in the study or put the subject at increased risk
* Intake of statins. If needed to obtain the recruitment goals, we will accept people using a low dose of statin. Simvastatin 10 mg or Pravastatin 10-20 mg will be accepted, but not higher doses or the drugs Lipitor/Atorvastatin and Crestor/Rosuvastatin.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in waist circumference in the CPH group as compared to placebo/casein at week 12 | At baseline visit and end visit (week 12)
  Waist circumference will be measured using anthropometric tape over light clothing. For waist circumference, the minimum circumference between the iliac crest and the rib cage will be used.

SECONDARY OUTCOMES:
Changes from baseline in glucagon-like peptide 1 (GLP-1, hormone involved in appetite and metabolism regulation) in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Measured in plasma using immunological methods (ELISA). All plasma samples will be kept on ice directly after collection, and relevant inhibitors will be added.
Changes from baseline in gastric inhibitory polypeptide (GIP, hormone involved in metabolism regulation) in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Measured in plasma using immunological methods (ELISA). All plasma samples will be kept on ice directly after collection, and relevant inhibitors will be added.
Changes from baseline in ghrelin (hormone involved in appetite regulation) in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Measured in plasma using immunological methods (ELISA). All plasma samples will be kept on ice directly after collection, and relevant inhibitors will be added.
Changes from baseline in heart rate in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  The heart rate will be registered after 5 minutes of supine rest using a Schiller BP-200
Changes from baseline in blood pressure in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  The blood pressure will be registered after 5 minutes of supine rest using a blood pressure monitor.
Changes from baseline in waist/hip ratio in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Waist and hip circumference will be measured using anthropometric tape over light clothing. For waist circumference, the minimum circumference between the iliac crest and the rib cage will be used. For hip circumference, the maximum measurement over the great trochanters will be used.
Changes from baseline in waist/height ratio in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Height will be measured with a wall-mounted stadiometer. Waist circumference will be measured using anthropometric tape over light clothing. The minimum circumference between the iliac crest and the rib cage will be used.
Changes from baseline in the Quick1 surrogate marker forinsulin sensitivity in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Glucose and insulin will be measured in serum by routine laboratories. Quick1 will be calculated by 1 / (log(fasting insulin μU/mL) + log(fasting glucose mg/dL)
Changes from baseline in serum glucose in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Changes from baseline in serum insulin c-peptide in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Changes from baseline in serum insulin in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Changes from baseline in serum total cholesterol in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Changes from baseline in serum triacylglycerol (TAG) in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Change from baseline in serum non-esterified fatty acids (NEFA) in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Change from baseline in serum non-HDL cholesterol in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Change from baseline in serum CRP in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Will be measured in serum by routine laboratories
Change from baseline in serum HDL cholesterol/LDL cholesterol size ratio in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Lipoprotein profile will be analysed by exclusion gel chromatography.
Change from baseline in serum ceramides in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  The ceramides in plasma will be analysed by LC-MS.
Change from baseline in fat mass/fat-free mass ratio in the CPH group as compared to placebo/casein | At baseline visit and end visit (week 12)
  Bioelectrical impedance measurement will be used for the assessment of body composition.
Changes in antioxidant capacity in the CPH group as compared to placebo/casein at week 12 | At baseline visit and end visit (week 12)
  Measured in plasma by a commercial kit (Sigma Aldrich, MAK187)
Changes in serum acetylcarnitine/palmitoylcarnitine ratio in the CPH group as compared to placebo/casein at week 12 | At baseline visit and end visit (week 12)
  Short-, medium-, and long-chain acylcarnitines, will be analysed in serum using LC/MS/MS.
Changes in serum octanoylcarnitine in the CPH group as compared to placebo/casein at week 12 | At baseline visit and end visit (week 12)
  Plasma choline, betaine, free carnitine and its precursors: trimethyllysine and γ-butyrobetaine, as well as short-, medium-, and long-chain acylcarnitines, will be analysed in serum using LC/MS/MS. Stable isotope dilution LC/MS/MS will be used for quantification of trimethylamine oxide (TMAO), dimethylglycine (DMG), choline and betaine. Plasma metabolites of the TCA cycle and amino acids-kynurenine-nicotinamide pathway will be measured by LC-MS.
Changes in serum TMAO (trimethylamine N-oxide) in the CPH group as compared to placebo/casein at week 12 | At baseline visit and end visit (week 12)
  Stable isotope dilution LC/MS/MS will be used for quantification of trimethylamine oxide (TMAO).
Changes from baseline in the serum anti-inflammatory fatty acid index in the CPH group as compared to placebo at Week 12. | At baseline visit and end visit (week 12)
  Fatty acid composition will be analysed using GC/MS. The anti-inflammatory fatty acid index is calculated as ((C22:5n-3 + C22:6n-3 + C20:3n-6 + C20:5n-3)/C20:4n-6)*100

CONTACTS AND LOCATIONS:
Overall Officials: Rolf K Berge, PhD, Study Director — University of Bergen, Norway
Locations (1):
- Research Unit for Health Trials, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No